CLINICAL TRIAL: NCT02777203
Title: Safety and Efficacy of Contained Electromechanical Power Morcellation Systems for Laparoscopic Hysterectomy and Myomectomy
Brief Title: Power Morcellation Systems for Laparoscopic Hysterectomy and Myomectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Espiner Medical LTD (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AHCIRB 6310 Power Morcellation
Record Dates: First submitted 2016-05-10; First posted 2016-05-19 (Estimated); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Leiomyoma
Keywords: morcellation; myomectomy; hysterectomy
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EcoSac 46 400 ECO-T morcellation bag cohort (Other): Prospective study of one cohort of subjects undergoing power morcellation within the EcoSac 46 400 ECO-T morcellation bag after a laparoscopic or robotic-assisted hysterectomy or myomectomy.
  Interventions: Device: EcoSac 400 ECO-T

INTERVENTIONS:
Device: EcoSac 400 ECO-T — Laparoscopy will be performed in the standard multi-port technique. The specimen will be morcellated in the EcoSac400 ECO-T bag. This study is a pilot study with one arm (all patients will use the new EcoSac400 ECO-T bag.

SUMMARY:
The purpose of this study is to determine the safety and efficacy of insufflated bags for electromechanical power morcellation during laparoscopic hysterectomy and myomectomy for tissue removal and to observe the integrity of the bags throughout and after insufflation and power morcellation.

The hypothesis is the bags will remain in tact without leakage from the bags during and after power morcellation using the described contained system, confirming the safety and efficacy of the systems.

DETAILED DESCRIPTION:
Uterine leiomyoma (fibroids) are non-cancerous smooth muscle tumors that can cause heavy menstrual bleeding, pain, and pressure. Common surgical treatment modalities are hysterectomy (removal of the uterus) or myomectomy (removal of the fibroid). Minimally invasive surgical techniques (laparoscopy) are generally recommended due to improved recovery time, decrease infection risk, decreased bleeding risk and overall decreased morbidity and mortality risks.

In order to remove a large uterus or large fibroids laparoscopically, a power morcellator is often used to cut the specimen into smaller pieces that can be removed through small incisions. Due to the concern regarding spread of small amounts of tissue during power morcellation, many surgeons are advocating contained power morcellation, i.e. morcellation inside a specimen bag.

This study will be evaluating the efficacy of contained morcellation using a specific specimen bag. Morcellation will be performed in the designated bag. The bag will then be removed evaluated for any egg albumin leakage. If there is no leakage, it can be inferred that there is no tissue is spread during the contained morcellation process using this bag.

ELIGIBILITY:
Inclusion Criteria:

* adult premenopausal women (equal or greater than 18 years old)
* no symptoms of menopause
* undergoing robotic or laparoscopic total or supracervical hysterectomies or myomectomies for the indication of symptomatic uterine fibroids
* not candidates for specimen removal via mini-laparotomy incision (as deemed by the study surgeon) or who have refused mini-laparotomy
* endometrial biopsy with no suspicion for malignancy

Exclusion Criteria:

* known or suspected malignancy
* peri- or post-menopausal women
* specimen that can be removed without power morcellation (e.g., vaginally or through laparoscopic trocars)
* adults unable to consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-05; Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Miller, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Advocate Lutheran General Hospital, Park Ridge, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cholkeri-Singh A, Miller CE. Power morcellation in a specimen bag. J Minim Invasive Gynecol. 2015 Feb;22(2):160. doi: 10.1016/j.jmig.2014.10.012. Epub 2014 Oct 18. PMID 25460317
- [Background] Cohen SL, Einarsson JI, Wang KC, Brown D, Boruta D, Scheib SA, Fader AN, Shibley T. Contained power morcellation within an insufflated isolation bag. Obstet Gynecol. 2014 Sep;124(3):491-497. doi: 10.1097/AOG.0000000000000421. PMID 25162248
- [Background] Einarsson JI, Cohen SL, Fuchs N, Wang KC. In-bag morcellation. J Minim Invasive Gynecol. 2014 Sep-Oct;21(5):951-3. doi: 10.1016/j.jmig.2014.04.010. Epub 2014 Apr 25. PMID 24769447
- [Background] Kho KA, Anderson TL, Nezhat CH. Intracorporeal electromechanical tissue morcellation: a critical review and recommendations for clinical practice. Obstet Gynecol. 2014 Oct;124(4):787-793. doi: 10.1097/AOG.0000000000000448. PMID 25198260
- [Background] Vargas MV, Cohen SL, Fuchs-Weizman N, Wang KC, Manoucheri E, Vitonis AF, Einarsson JI. Open power morcellation versus contained power morcellation within an insufflated isolation bag: comparison of perioperative outcomes. J Minim Invasive Gynecol. 2015 Mar-Apr;22(3):433-8. doi: 10.1016/j.jmig.2014.11.010. Epub 2014 Nov 29. PMID 25452122

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Undergoing Myomectomy or Hysterectomy With Morcellation: Subjects undergoing power morcellation with the EcoSac 400 ECO-T morcellation bag after a laparoscopic or robotic-assisted hysterectomy or myomectomy.
Period: Overall Study
Arm/Group | Patients Undergoing Myomectomy or Hysterectomy With Morcellation
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: women who underwent laparoscopic surgery utilizing morcellation in a bag
Groups:
- Only One Arm Was Utilized: one arm
Arm/Group | Only One Arm Was Utilized
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 60
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 53
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 14
  White | 43
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Egg Albumin Leakage.
Description: After morcellation is complete, the bag was removed from the abdomen and taken out of the operating room to the frozen section room to inspect the integrity of the bag. Five hundred milliliters of egg albumin combined with 0.5 milliliters of methylene blue were placed into the bag to assess for any leakage.Visual inspection will be used to assess leakage from the bag with outcome measures of "yes" or "no."
Time Frame: Day 0 through the end of morcellation, approximately 30 minutes.
Measure: Count of Participants; unit: Participants
Groups:
- Patients Utilizing EcosacT400 Bag: Patients undergoing hysterectomy and myomectomy utilizing morcellation and new EcosacT400 bag
Arm/Group | Patients Utilizing EcosacT400 Bag
Number analyzed (Participants) | 60
Participants | 0

2. Secondary Outcome: Morcellation Time
Description: Time (in minutes) from insertion of the bag to removal of the bag
Time Frame: Day 0 through the end of morcellation, approximately 30 minutes.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Patients Utilizing EcosacT400 Bag: Patients undergoing hysterectomy and myomectomy utilizing morcellation and EcosacT400 bag
Arm/Group | Patients Utilizing EcosacT400 Bag
Number analyzed (Participants) | 60
minutes | 26.3 (14.6)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Patient were followed continuously for six weeks post-operatively.
Groups:
- Patients Utilizing ecosacT400 Bag: Patients undergoing hysterectomy and myomectomy utilizing morcellation and the EcosacT400 bag
Arm/Group | Patients Utilizing ecosacT400 Bag
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 25/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Utilizing ecosacT400 Bag (N=60)
post op urinary retention (Renal and urinary disorders) | 3 (3) — post operative urinary retention
umbillical drainage (Surgical and medical procedures) | 5 (5) — Incisional drainage post operative ( from surgical site)
Incisional pain (Surgical and medical procedures) | 1 (1) — post operative incisional pain
chest pain (Surgical and medical procedures) | 2 (2) — Post operative chest pain due to Co2 gas
diarrhea (Gastrointestinal disorders) | 3 (3) — Post operative diarrhea related to antibiotic use
back pain (Musculoskeletal and connective tissue disorders) | 1 (1) — post operative back pain
Fever (Infections and infestations) | 2 (2) — Post operative fever
leg numbness (Nervous system disorders) | 1 (1) — Post operative numbness in thigh due to lithotomy positioning
Broken instrument (Surgical and medical procedures) | 1 (1) — A surgical instrument used during surgery broke apart inside patient .Surgery was stopped and all pieces were removed
bruising around incision sites (Surgical and medical procedures) | 1 (1) — Bruising noted around incisions
post operative nausea (Gastrointestinal disorders) | 1 (1) — nausea after surgery lasting greater than 24 hours
Fatigue (Surgical and medical procedures) | 1 (1) — Fatigue after surgery
rash (Skin and subcutaneous tissue disorders) | 1 (1) — Post operative rash
Peritoneal rent (Injury, poisoning and procedural complications) | 1 (1) — Espiner bag was introduced through umbilical port while not under direct vision and a rent was made in the peritoneum. the area was explored and no issues noted
constipation (Gastrointestinal disorders) | 1 (1) — post operative constipation
Vaginal discharge/yeast infection (Surgical and medical procedures) | 2 (2) — vaginal discharge/yeast infection post operative associated with antibiotic use

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-04-11): https://cdn.clinicaltrials.gov/large-docs/03/NCT02777203/Prot_SAP_000.pdf
  • Informed Consent Form (2017-07-05): https://cdn.clinicaltrials.gov/large-docs/03/NCT02777203/ICF_001.pdf